CLINICAL TRIAL: NCT01292473
Title: A Phase III, Multicenter, Randomized, Double-blind, Dose-ranging, Placebo-controlled Study to Evaluate the Efficacy, Response Duration and Safety of Xolair (Omalizumab) in Patients With Chronic Idiopathic Urticaria (CIU)/Chronic Spontaneous Urticaria Who Remain Symptomatic Despite Antihistamine Treatment (H1)
Brief Title: A Study to Evaluate the Efficacy, Response Duration and Safety of Xolair (Omalizumab) in Patients With Chronic Idiopathic Urticaria (CIU)/Chronic Spontaneous Urticaria (CSU) Who Remain Symptomatic Despite Antihistamine Treatment (H1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Q4882g
Record Dates: First submitted 2011-02-07; First posted 2011-02-09 (Estimated); Results first posted 2013-09-02 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Idiopathic Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Experimental): Placebo subcutaneously (sc) every 4 weeks
  Interventions: Drug: Placebo; Drug: Omalizumab
- Omalizumab 75 mg (Experimental): Omalizumab 75 mg sc every 4 weeks
  Interventions: Drug: Omalizumab
- Omalizumab 150 mg (Experimental): Omalizumab 150 mg sc every 4 weeks
  Interventions: Drug: Omalizumab
- Omalizumab 300 mg (Experimental): Omalizumab 300 mg sc every 4 weeks.
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Placebo — Placebo was supplied lyophilized in vials.
  Arms: Placebo
Drug: Omalizumab — Omalizumab was supplied lyophilized in vials.
  Other Names: Xolair

SUMMARY:
The study is a global Phase III, multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of omalizumab administered subcutaneously as an add-on therapy for the treatment of adolescent and adult patients aged 12-75 who have been diagnosed with refractory CIU and who remain symptomatic despite standard-dosed H1 antihistamine treatment.

DETAILED DESCRIPTION:
The trial incorporated a Type I error control plan, as follows:

The testing of the primary endpoint was conducted in the following hierarchical order. A p-value that is less than 0.05 can only be claimed statistically significant if statistical significance has been claimed at the previous stage.

* Stage 1: Omalizumab 300-mg group vs. placebo
* Stage 2: Omalizumab 150-mg group vs. placebo
* Stage 3: Omalizumab 75-mg group vs. placebo

A hierarchical analysis of the secondary endpoints was performed for each dose found to be significant in the primary endpoint. A p-value that is less than 0.05 can only be claimed statistically significant if statistical significance has been claimed at the previous stage.

* Stage 1: Change from baseline in Urticaria Activity Score (UAS7) at Week 12
* Stage 2: Change from baseline in the weekly number of hives score at Week 12
* Stage 3: Time to weekly itch severity score Minimally Important Difference (MID) response at Week 12
* Stage 4: Proportion of patients with UAS7 ≤ 6 at Week 12
* Stage 5: Proportion of weekly itch severity score MID Responders at Week 12
* Stage 6: Change from baseline in weekly size of the largest hive score at Week 12
* Stage 7: Change from baseline in overall Dermatology Life Quality Index (DLQI) score at Week 12
* Stage 8: Proportion of angioedema-free days from Week 4 to Week 12

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic Idiopathic Urticaria (CIU)/Chronic Spontaneous Urticaria (CSU) CIU/CSU refractory to H1 antihistamines at the time of randomization.

Exclusion Criteria:

* Treatment with an investigational agent within 30 days prior to screening.
* Weight < 20 kg (44 lbs).
* Clearly defined underlying etiology for chronic urticarias other than CIU.
* Evidence of parasitic infection.
* Atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus, or other skin disease associated with itch.
* Previous treatment with omalizumab within a year prior to screening.
* Routine doses of the following medications within 30 days prior to screening: Systemic or cutaneous (topical) corticosteroids (prescription or over the counter), hydroxychloroquine, methotrexate, cyclosporine, or cyclophosphamide.
* Intravenous (IV) immunoglobulin G (IVIG), or plasmapheresis within 30 days prior to screening.
* Regular (daily/every other day) doxepin (oral) use within 6 weeks prior to screening.
* Any H2 antihistamine use within 7 days prior to screening.
* Any leukotriene receptor antagonist (LTRA) (montelukast or zafirlukast) within 7 days prior to screening.
* Any H1 antihistamines at greater than approved doses within 3 days prior to screening.
* Patients with current malignancy, history of malignancy, or currently under work-up for suspected malignancy except non-melanoma skin cancer that has been treated or excised and is considered resolved.
* Hypersensitivity to omalizumab or any component of the formulation.
* History of anaphylactic shock.
* Presence of clinically significant cardiovascular, neurological, psychiatric, metabolic, or other pathological conditions that could interfere with the interpretation of the study results and or compromise the safety of the patients.
* Evidence of current drug or alcohol abuse.
* Nursing women or women of childbearing potential, unless they meet the following definition of post-menopausal: 12 months of natural amenorrhea or 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone (FSH) levels > 40 milli-international units per milliliter (mIU/mL) or 6 weeks post surgical bilateral oophorectomy (with or without hysterectomy) or hysterectomy or are using one or more of the following acceptable methods of contraception: surgical sterilization, hormonal contraception, and double-barrier methods.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin E Rosén, MD, PhD, Study Director — Genentech, Inc.
Locations (58):
- United States (34):
  - La Jolla, California
  - Los Angeles, California
  - Redwood City, California
  - Walnut Creek, California
  - Denver, Colorado
  - Miami, Florida
  - Savannah, Georgia
  - Woodstock, Georgia
  - Shiloh, Illinois
  - Indianapolis, Indiana
  - Overland Park, Kansas
  - Baltimore, Maryland
  - Wheaton, Maryland
  - Ypsilanti, Michigan
  - Omaha, Nebraska
  - Brick, New Jersey
  - Bayside, New York
  - Brooklyn, New York
  - North Syracuse, New York
  - Rochester, New York
  - Rockville Centre, New York
  - The Bronx, New York
  - Asheville, North Carolina
  - Canton, Ohio
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - El Paso, Texas
  - Sandy City, Utah
  - Seattle, Washington
  - Spokane, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Denmark (2):
  - Aarhus
  - Copenhagen
- France (3):
  - Montpellier
  - Nice
  - Paris
- Germany (6):
  - Bonn
  - Hanover
  - Leipzig
  - Mainz
  - München
  - Münster
- Italy (2):
  - Genova
  - Milan
- Poland (5):
  - Gdansk
  - Krakow
  - Lodz
  - Warsaw
  - Wroclaw
- Spain (2):
  - Barcelona
  - Madrid
- Turkey (Türkiye) (4):
  - Ankara
  - Istanbul
  - Izmir
  - Kayseri

REFERENCES:
- [Derived] Casale TB, Trzaskoma B, Holden M, Bernstein JA, Maurer M. Does angioedema in patients with chronic spontaneous urticaria impact response to omalizumab? World Allergy Organ J. 2024 Aug 5;17(8):100943. doi: 10.1016/j.waojou.2024.100943. eCollection 2024 Aug. PMID 39193419
- [Derived] Ferrer M, Gimenez-Arnau A, Saldana D, Janssens N, Balp MM, Khalil S, Risson V. Predicting Chronic Spontaneous Urticaria Symptom Return After Omalizumab Treatment Discontinuation: Exploratory Analysis. J Allergy Clin Immunol Pract. 2018 Jul-Aug;6(4):1191-1197.e5. doi: 10.1016/j.jaip.2018.04.003. Epub 2018 Apr 12. PMID 29655772
- [Derived] Goldstein S, Gabriel S, Kianifard F, Ortiz B, Skoner DP. Clinical features of adolescents with chronic idiopathic or spontaneous urticaria: Review of omalizumab clinical trials. Ann Allergy Asthma Immunol. 2017 Apr;118(4):500-504. doi: 10.1016/j.anai.2017.02.003. PMID 28390587
- [Derived] Saini SS, Omachi TA, Trzaskoma B, Hulter HN, Rosen K, Sterba PM, Courneya JP, Lackey A, Chen H. Effect of Omalizumab on Blood Basophil Counts in Patients with Chronic Idiopathic/Spontaneous Urticaria. J Invest Dermatol. 2017 Apr;137(4):958-961. doi: 10.1016/j.jid.2016.11.025. Epub 2016 Dec 6. No abstract available. PMID 27939380
- [Derived] Gimenez-Arnau AM, Spector S, Antonova E, Trzaskoma B, Rosen K, Omachi TA, Stull D, Balp MM, Murphy T. Improvement of sleep in patients with chronic idiopathic/spontaneous urticaria treated with omalizumab: results of three randomized, double-blind, placebo-controlled studies. Clin Transl Allergy. 2016 Aug 18;6:32. doi: 10.1186/s13601-016-0120-0. eCollection 2016. PMID 27540466
- [Derived] Zazzali JL, Kaplan A, Maurer M, Raimundo K, Trzaskoma B, Solari PG, Antonova E, Mendelson M, Rosen KE. Angioedema in the omalizumab chronic idiopathic/spontaneous urticaria pivotal studies. Ann Allergy Asthma Immunol. 2016 Oct;117(4):370-377.e1. doi: 10.1016/j.anai.2016.06.024. Epub 2016 Jul 14. PMID 27424128
- [Derived] Casale TB, Bernstein JA, Maurer M, Saini SS, Trzaskoma B, Chen H, Grattan CE, Gimenez-Arnau A, Kaplan AP, Rosen K. Similar Efficacy with Omalizumab in Chronic Idiopathic/Spontaneous Urticaria Despite Different Background Therapy. J Allergy Clin Immunol Pract. 2015 Sep-Oct;3(5):743-50.e1. doi: 10.1016/j.jaip.2015.04.015. Epub 2015 Jun 6. PMID 26054553
- [Derived] Maurer M, Rosen K, Hsieh HJ, Saini S, Grattan C, Gimenez-Arnau A, Agarwal S, Doyle R, Canvin J, Kaplan A, Casale T. Omalizumab for the treatment of chronic idiopathic or spontaneous urticaria. N Engl J Med. 2013 Mar 7;368(10):924-35. doi: 10.1056/NEJMoa1215372. Epub 2013 Feb 24. PMID 23432142

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Started | 79 | 82 | 83 | 79
Completed | 74 | 75 | 74 | 67
Not Completed | 5 | 7 | 9 | 12
Not completed — Adverse Event | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 3 | 4 | 3 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Disease Progression | 0 | 1 | 3 | 6

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat population: All randomized patients who received at least one dose of study drug.
Groups:
- Placebo: Placebo administered subcutaneously (sc) every 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg | Total
Number analyzed (Participants) | 79 | 82 | 82 | 79 | 322
Age Continuous [Mean (Standard Deviation); unit: Years] | 43.1 (12.5) | 39.7 (15.0) | 43.0 (13.2) | 44.3 (13.7) | 42.5 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 61 | 65 | 63 | 244
  Male | 24 | 21 | 17 | 16 | 78

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Weekly Itch Severity Score at Week 12
Description: The weekly itch severity score is the sum of the daily itch severity scores over 7 days and ranges from 0 to 21. The daily itch severity score is the average of the morning and evening scores on a scale of 0 (none) to 3 (severe). The Baseline weekly itch severity score is the sum of the daily itch severity scores over the 7 days prior to the first treatment. A higher itch severity score indicates more severe itching. A negative change score indicates improvement.
Time Frame: Baseline, Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 79 | 82 | 82 | 79
Units on a scale | -5.14 (5.58) | -5.87 (6.45) | -8.14 (6.44) | -9.77 (5.95)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 75 mg groups; Test type: Superiority or Other; p = 0.4637, ANCOVA — Refer to the Type-I error control plan; Covariates included in the analysis were baseline weekly itch severity score (< 13 vs ≥ 13) and baseline weight (< 80 kg vs ≥ 80 kg); Least Squares Mean Difference = -0.69, 95% CI 2-sided [-2.54 to 1.16]
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 150 mg groups; Test type: Superiority or Other; p = 0.0011, ANCOVA — Refer to the Type-I error control plan; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -3.04, 95% CI 2-sided [-4.85 to -1.24]
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — Refer to the Type-I error control plan; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -4.81, 95% CI 2-sided [-6.49 to -3.13]

2. Secondary Outcome: Change From Baseline in the Weekly Urticaria Activity Score (UAS7) at Week 12
Description: The urticaria activity score (UAS) is a composite of scores on a scale of 0 (none) to 3 (intense/severe) for 1) the number of wheals (hives); and 2) the intensity of the itch, measured twice daily (morning and evening). Daily UAS is the average of morning and evening scores (ranging from 0-6) and the UAS7 is the sum of the daily UAS over 7 days (ranging from 0-42). Baseline UAS7 is calculated using data from the 7 days prior to the first treatment date. A higher UAS indicates more urticaria activity. A negative change score indicates improvement.
Time Frame: Baseline, Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 79 | 82 | 82 | 79
Units on a scale | -10.36 (11.61) | -13.08 (12.67) | -17.89 (13.23) | -21.74 (12.78)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 75 mg groups; Test type: Superiority or Other; p = 0.1575, ANCOVA — Refer to the Type-I error control plan. The p-value was not evaluated for statistical significance in accordance with the Type I error control plan provided in the Detailed Description; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg); Least Squares Mean Difference = -2.73, 95% CI 2-sided [-6.53 to 1.07]
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 150 mg groups; Test type: Superiority or Other; p = 0.0001, ANCOVA — Refer to the Type-I error control plan; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg); Least Squares Mean Difference = -7.69, 95% CI [-11.49 to -3.88]
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — Refer to the Type-I error control plan; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg); Least Squares Mean Difference = -12.40, 95% CI 2-sided [-16.13 to -8.66]

3. Secondary Outcome: Change From Baseline in the Weekly Number of Hives Score at Week 12
Description: The weekly hives score is the sum of the daily hives scores over 7 days and ranges from 0 to 21. The number of hives is measured twice daily (morning and evening) on a scale of 0 (none) to 3 (> 12 hives per 12 hours). The daily hives score is the average of the morning and evening scores. The Baseline score is the sum of the daily hives scores over the 7 days prior to the first treatment. A higher score indicates more hives. A negative change score indicates improvement.
Time Frame: Baseline, Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 79 | 82 | 82 | 79
Units on a scale | -5.22 (6.56) | -7.21 (6.96) | -9.75 (7.28) | -11.97 (7.58)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 75 mg groups; Test type: Superiority or Other; p = 0.0603, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Covariates included in the analysis were baseline weekly number of hives (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg); Least Squares Mean Difference = -2.01, 95% CI 2-sided [-4.11 to 0.09]
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 150 mg groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — Refer to the Type-I error control plan; [statistical method as in outcome 3, analysis 1]; Least Squares Mean Difference = -4.51, 95% CI 2-sided [-6.65 to -2.36]
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — Refer to the Type-I error control plan; [statistical method as in outcome 3, analysis 1]; Least Squares Mean Difference = -7.09, 95% CI 2-sided [-9.26 to -4.93]

4. Secondary Outcome: Time to Minimally Important Difference (MID) Response in the Weekly Itch Severity Score by Week 12
Description: The weekly itch severity score is the sum of the daily itch severity scores over 7 days and ranges from 0 to 21. The daily itch severity score is the average of the morning and evening scores on a scale of 0 (none) to 3 (severe). The Baseline weekly itch severity score is the sum of the daily itch severity scores over the 7 days prior to the first treatment. A higher itch severity score indicates more severe itching. A negative change score indicates improvement.
  The MID response for weekly itch severity score was defined as a reduction from baseline in weekly itch severity score of 5 points or more. The time to weekly itch severity score MID response was defined as the time (in weeks) from Day 1 to the study week when weekly itch severity score MID response was first achieved.
Time Frame: by Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 79 | 82 | 82 | 79
Weeks | 4.0 [3.0 to 5.0] | 2.0 [2.0 to 3.0] | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; The null hypothesis is that there is no difference between Placebo and Omalizumab 75 mg; Test type: Superiority or Other; p = 0.0478, Cox proportional hazards model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [1.00 to 2.05]
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 150 mg groups; Test type: Superiority or Other; p = 0.0101, Cox proportional hazards model — Refer to the Type-I error control plan; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.59, 95% CI 2-sided [1.12 to 2.26]
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis is that there is no difference between placebo and omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, Cox proportional hazards model — Refer to the Type-I error control plan; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 2.12, 95% CI 2-sided [1.48 to 3.03]

5. Secondary Outcome: Percentage of Participants With a UAS7 Less Than or Equal to 6 at Week 12
Description: as for outcome 2
Time Frame: Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 79 | 82 | 82 | 79
Percentage of participants | 19.0 | 26.8 | 42.7 | 65.8
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 75 mg groups; Test type: Superiority or Other; p = 0.3419, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg)
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 150 mg groups; Test type: Superiority or Other; p = 0.0010, Cochran-Mantel-Haenszel — Refer to the Type-I error control plan; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg)
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis is that there is no difference between placebo and omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Refer to the Type-I error control plan; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg)

6. Secondary Outcome: Percentage of Weekly Itch Severity Score MID Responders at Week 12
Description: The weekly itch severity score is the sum of the daily itch severity scores over 7 days and ranges from 0 to 21. The daily itch severity score is the average of the morning and evening scores on a scale of 0 (none) to 3 (severe). The Baseline weekly itch severity score is the sum of the daily itch severity scores over the 7 days prior to the first treatment. A higher itch severity score indicates more severe itching. A negative change score indicates improvement.
  The MID response for weekly itch severity score was defined as a reduction from baseline in weekly itch severity score of 5 points or more. This outcome measure shows the percentage of participants classified as MID Responders at Week 12, meaning their weekly itch severity scores at Week 12 were at least 5 points lower than at Baseline.
Time Frame: Baseline, Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 79 | 82 | 82 | 79
Percentage of participants | 48.1 | 56.1 | 69.5 | 78.5
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 75 mg groups; Test type: Superiority or Other; p = 0.4366, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 150 mg groups; Test type: Superiority or Other; p = 0.0045, Cochran-Mantel-Haenszel — Refer to the Type-I error control plan; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Refer to the Type-I error control plan; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in the Weekly Size of the Largest Hive Score at Week 12
Description: The size of the largest hive is assessed twice daily (morning and evening) on a scale of 0 (none) to 3 (> 2.5 cm). The daily score is the average of the morning and evening scores. The weekly size of the largest hive score is the sum of the daily scores over 7 days, and ranges from 0 to 21. The Baseline weekly size of the largest hive score is the sum of daily scores over the 7 days prior to the first treatment. A higher score indicates larger hives. A negative change score indicates a reduction in hive size.
Time Frame: Baseline, Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 79 | 82 | 82 | 79
Units on a scale | -4.04 (5.55) [-18.5 to 7.5] | -6.52 (6.33) [-5.61 to -1.90] | -7.84 (6.75) [-12.61 to -9.39] | -11.00 (7.18)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 75 mg groups; Test type: Superiority or Other; p = 0.0082, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Covariates included in the analysis were baseline weekly size of largest hive score (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg); Least Squares Mean Difference = -2.48, 95% CI 2-sided [-4.32 to -0.65]
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 150 mg groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — Refer to the Type-I error control plan; [statistical method as in outcome 7, analysis 1]; Least Squares Mean Difference = -3.76, 95% CI 2-sided [-5.61 to -1.90]
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis is that there is no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — Refer to the Type-I error control plan; [statistical method as in outcome 7, analysis 1]; Least Squares Mean Difference = -7.15, 95% CI 2-sided [-9.03 to -5.27]

8. Secondary Outcome: Change From Baseline in the Overall Dermatology Life Quality Index (DLQI) at Week 12
Description: The dermatology life quality index (DLQI) is a 10-item dermatology-specific health-related quality of life measure. Participants rate their dermatology symptoms as well as the impact of their skin condition on various aspects of their lives on a scale of 0 (Not at all) to 3 (Very much). The overall DLQI is the sum of the responses to the 10 items and ranges from 0 to 30. A lower score indicates a better quality of life. A negative change score indicates improvement.
Time Frame: Baseline, Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least one dose of study drug and who had a DLQI score at Week 12.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 69 | 68 | 70 | 73
Units on a scale | -6.09 (7.47) | -7.50 (7.16) | -8.29 (6.31) | -10.15 (6.83)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 75 mg groups; Test type: Superiority or Other; p = 0.1207, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Covariates included in the analysis were baseline overall DLQI score (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg); Least Squares Mean Difference = -1.68, 95% CI 2-sided [-3.82 to 0.45]
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 150 mg groups; Test type: Superiority or Other; p = 0.0215, ANCOVA — Refer to the Type-I error control plan; [statistical method as in outcome 8, analysis 1]; Least Squares Mean Difference = -2.51, 95% CI 2-sided [-4.64 to -0.38]
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 300 mg groups; Test type: Superiority or Other; p = 0.0004, ANCOVA — Refer to the Type-I error control plan; [statistical method as in outcome 8, analysis 1]; Least Squares Mean Difference = -3.79, 95% CI 2-sided [-5.85 to -1.73]

9. Secondary Outcome: Percentage of Angioedema-free Days From Week 4 to Week 12
Description: The percentage of angioedema-free days from Weeks 4 to 12 was defined as the number of days a patient reported as angioedema-free in the daily diary divided by the total number of days with a non-missing diary entry, starting at the Week 4 visit and ending the day prior to the Week 12 visit.
Time Frame: Week 4 to Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least one dose of study drug. Patients who withdrew before the Week 4 visit or who had missing responses for more than 40% of the daily diary entries between the Week 4 visit and the Week 12 visit were not included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 70 | 71 | 74 | 74
Percentage of days | 89.2 (19.0) | 93.5 (14.9) | 91.6 (17.4) | 95.5 (14.5)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 75 mg groups; Test type: Superiority or Other; p = 0.1361, Stratified Wilcoxon — [p-value comment as in outcome 2, analysis 1]; Stratification variables included in the analysis were presence of angioedema at baseline (yes vs no) and baseline weight (< 80 kg vs ≥ 80 kg)
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 150 mg groups; Test type: Superiority or Other; p = 0.0905, Stratified Wilcoxon — Refer to the Type-I error control plan; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis is that there is no difference between the placebo and omalizumab 300 mg; Test type: Superiority or Other; p < 0.0001, Stratified Wilcoxon — Refer to the Type-I error control plan; [statistical method as in outcome 9, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of first treatment through the end of the study (up to 28 weeks).
Description: Safety evaluable set: All randomized participants who received at least one dose of study drug. Data are presented according to the doses actually received - one subject randomized to the 150 mg group withdrew before dosing, and six subjects randomized to the 75 mg group actually received 150 mg.
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Serious Adverse Events (participants affected / at risk) | 2/79 | 1/76 | 1/88 | 5/79
Other Adverse Events (participants affected / at risk) | 35/79 | 30/76 | 42/88 | 35/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=79) | Omalizumab 75 mg (N=76) | Omalizumab 150 mg (N=88) | Omalizumab 300 mg (N=79)
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Tonsillectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Malignant melanoma in situ (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=79) | Omalizumab 75 mg (N=76) | Omalizumab 150 mg (N=88) | Omalizumab 300 mg (N=79)
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 4 | 3
Nasopharyngitis (Infections and infestations) | 15 | 13 | 15 | 12
Upper respiratory tract infection (Infections and infestations) | 7 | 0 | 2 | 6
Influenza (Infections and infestations) | 4 | 5 | 3 | 2
Sinusitis (Infections and infestations) | 2 | 3 | 2 | 6
Bronchitis (Infections and infestations) | 2 | 4 | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 4 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 4
Headache (Nervous system disorders) | 7 | 4 | 18 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2 | 2
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 3 | 8 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.